CLINICAL TRIAL: NCT04703504
Title: RAndomized Controlled Trial of a Multiple INtervention proGram to Decrease Heart Failure Rehospitalization
Acronym: RACING-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment targets will not be met
Sponsor: French Cardiology Society (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-06
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Decompensation
Keywords: heart failure; multiple intervention program
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multi-intervention (Experimental): * Automatic creation of discharge prescription (personalized checklist of possible therapeutic optimizations generated from clinical data entered into the platform. This checklist will comply with the recommendations on altered left ventricular ejection fraction from European Society of Cardiology 2016.
  * Automatic creation of documents for patient:
    * Reminder letter to make an appointment with his general practitioner (at 7 days) and cardiologist (1 month) and to report the prescribed blood test.
    * Drug prescription.
    * Prescription for blood tests (5 days and 25 days before seeing the general practitioner and cardiologist).
    * Therapeutic education documents
  * Patients will receive numerous messages (SMS / e-mail) in order to 1 / not forget their medical appointments, 2 / not to forget to make and bring back their blood test for the consultation, 3 / to perfect the therapeutic education advice provided previously
  Interventions: Other: Multiple intervention program
- Control (No Intervention): Discharge prescription according to the investigator's habits.

INTERVENTIONS:
Other: Multiple intervention program — Support for patient follow-up assisted by a computer program
  Arms: multi-intervention

SUMMARY:
The prevalence of heart failure (HF) is constantly increasing in France due to the aging of the population, better management of etiological factors and improved treatments (drug / interventional). On the other hand, re-hospitalizations for heart failure continue to increase, exceeding reception capacities and constitute a real challenge for current public health systems. The PRADO system provides administrative support (through a health insurance advisor) in the management of patient appointments with their doctors as well as home visits by a nurse trained in heart failure. Other interventional medical and educational interventions performed during an out-of-hospital consultation guided by a computer platform would help to optimize the care and continuity of care.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate the value of a multiple intervention program in reducing early readmissions for heat failure in patients hospitalized for cardiac decompensation.

This work will create an interventional assistance program to structure the exit consultation in order to optimize treatment, educate patients, ensure the continuity of hospital-city care and improve compliance (reminders) to reduce re-hospitalizations. This program will be carried out by using a computer platform allowing the systematization of output documents and the sending of messages (e-mail / SMS) for making appointments (medical consultations, biologicals sampling) and perfect therapeutic education.

ELIGIBILITY:
Inclusion Criteria:

* Heart decompensation requiring hospitalization and the use of intravenous diuretic therapy
* Left Ventricular Ejection Fraction ≤ 40%.

Exclusion Criteria:

* Hospitalization for cardiac decompensation leading to an invasive procedure (valve, coronary, etc.).
* Acute reversible cause of heart failure.
* Incurable disease (other than heart failure) or estimated life expectancy of less than one year.
* Patient transferred directly to another department or cardiac rehabilitation center.
* Significant cognitive impairment.
* Patient without cell phone or email.
* Linguistic or psychic refusal or inability to sign the informed consent.
* Current participation in a clinical tria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with a re-hospitalization due to heart decompensation | 3 months
  Defined as occurence of the need for hospitalization for cardiac decompensation justifying the use of intravenous diuretic therapy.

SECONDARY OUTCOMES:
Number of participants with a re-hospitalization due to heart decompensation | 12 months
  Defined as occurence of the need for hospitalization for cardiac decompensation justifying the use of intravenous diuretic therapy.
Number of re-hospitalization due to heart decompensation per patient | 12 months
  Defined as total number of hospitalization for heart decompensation during 1 year
Delay between discharge and re-hospitalization due to heart decompensation | 12 months
  Defined as time to first occurrence of re-hospitalization due to heart decompensation
Number of participants with death | 3 months
Number of participants with death | 12 months
Rate of pacemaker implantation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud GALAT, MD, Principal Investigator — CHU Henri Mondor, Créteil
Locations (8):
- France (8):
  - Hôpital Paul d'Egine, Champigny-sur-Marne
  - Hôpital Henri Mondor, Créteil
  - Hôpital Simone Veil, Eaubonne
  - Hôpitaux Nord-Ouest de Villefranche, Gleizé
  - Hôpital Européen Georges Pompidou, Paris
  - Polyclinique de Poitiers, Poitiers
  - Centre Cardiologique du Nord, Saint-Denis
  - Centre Hopsitalier Lucie et Raymond Aubrac, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No